CLINICAL TRIAL: NCT05824156
Title: Phase 2A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of CM-101 in Patients With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: CM-101 in NASH Patients - The SPLASH Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-NASH-201
Record Dates: First submitted 2021-12-06; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Anti-fibrotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 mg/kg CM-101 (Experimental): Subcutaneous injection CM-101 every 2 weeks
  Interventions: Biological: 5 mg/kg CM-101
- Placebo (Placebo Comparator): Subcutaneous Injection Placebo every 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 5 mg/kg CM-101 — CM-101, Monoclonal Ab blocking CCL24
  Arms: 5 mg/kg CM-101
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This phase 2a study is a multi-center, double-blind randomized, placebo-controlled study. The study is designed to determine the safety and tolerability of the anti-human CCL24 monoclonal antibody CM-101 in adult patients with non-cirrhotic nonalcoholic steatohepatitis (NASH) patients with stage 1c, 2 or 3 fibrosis. The patients will be randomized to 1 of 2 treatment groups: 5 mg/kg CM-101 or placebo.

DETAILED DESCRIPTION:
This study will consist of screening period, treatment period and follow-up period. Adults with NASH will be included. Each subject will undergo screening procedures within up to 42 days prior to Randomization, to assess eligibility to participate in the study. After randomization patients will receive a dose of investigational product once every 2 weeks for a total of 8 administrations. This will result in a total coverage of 16 weeks. Study participation will last for up to approximately 26 weeks (up to 6 weeks for screening followed by 14 weeks treatment and 6 weeks follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of steatohepatitis and fibrosis without cirrhosis on a diagnostic liver biopsy obtained within the 18 months prior to the start of treatment, and/or during the screening period with:

  a. NAS ≥ 4 with a score of at least 1 for each component (steatosis, ballooning degeneration and lobular inflammation) and b. Hepatic fibrosis stage F1c, 2 or 3 as defined by the NASH CRN scoring scale. F1c subjectspatients must have either: PRO-C3 >14 ng/ml or Liver stiffness value of >8.0 kPa measured by transient elastography
* Patients with presence of greater than or equals to (≥) 10 percent (%) steatosis on MRI-derived proton-density fat-fraction (PDFF) performed as part of the screening procedure or within 12 weeks prior to randomization
* Confirmation of disease status from time of biopsy by Transient Elastography performed during the screening period with liver stiffness value of 7-12 kPa.
* Patients with presence of ≥1 of the following risk factors:

  1. Obesity (BMI ≥30 kg/m2),
  2. Type 2 diabetes diagnosed per 2013 American Diabetes Association criteria,
  3. HTN per 2017 AHA Guidelines for Hypertension,
  4. ALT >1.5× upper limit of normal (ULN)
* Patients with a stable body mass index (BMI) between 25- 45 kg/m², both inclusive. Body weight is required to be stable (i.e., not varying by > 5% for at least 12 weeks) prior to study entry;
* Patients on chronic medication must be on a stable regimen for ≥ 12 weeks prior to Randomization and should attempt to maintain a stable dosing regimen during the study period;
* Patients must have the following laboratory parameters at screening:

  1. Total bilirubin < 1.5 mg/dL (26 micromol/L)
  2. AST < 5 x ULN
  3. INR < 1.3
  4. Creatinine clearance ≥60 mL/min as calculated by Cockcroft Gault equation;
  5. Alpha-fetoprotein in normal range (i.e. <20 ng/mL). If greater than normal, the patient requires a negative ultrasound for hepatocellular carcinoma within 12 weeks prior to randomization
* Women of childbearing potential must agree to use an approved form of contraception (e.g. oral, transdermal patch, implanted contraceptives, intrauterine device, diaphragm, condom, abstinence or surgical sterility) prior to randomization and for the duration of study participation through to 60 days after the last dose of the study medication. Confirmation that female patients are not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for documented postmenopausal or surgically sterilized women;
* Male patients must agree to use a barrier method of contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide) or abstinence for the duration of study participation through 60 days after the last dose of the study medication.
* Patients able to understand and sign a written informed consent form (ICF), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

* Patients with medical/surgical history of bariatric surgery procedures or bariatric device insertion or patients that are planned for such interventions;
* Patients taking weight loss medications;
* Evidence of drug induced steatohepatitis secondary to amiodarone, corticosteroids, estrogens, methotrexate, tetracycline, or other medications known to cause hepatic steatosis;
* History or presence of cirrhosis (compensated or decompensated) determined by histology or relevant medical complications and laboratory parameters;
* Model for End-stage Liver Disease (MELD) score >12;
* History of liver transplant, or current evaluation for or placement on a liver transplant waiting list;
* Abnormal laboratory screening values:

  1. Hemoglobin < 12.0 g/dL in males and < 11.0 g/dL in females
  2. Platelet count < 140,000/mm3
  3. Total white blood cells (WBC) < 3,000 cells/mm3
  4. Absolute neutrophil count (ANC) < 1,500 cells/mm3
  5. Serum albumin < 3.5 g/dL
* Screening ECG demonstrating prolongation of QT interval corrected by Fredericia Correction Formula (QTcF) of > 500 msec, or a history of clinically significant arrythmias
* History of other chronic liver diseases including:

  1. Alcoholic liver disease
  2. Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
  3. Hepatitis C as defined by presence of hepatitis C virus antibody (HCV-Ab) even if successfully treated with an antiviral regimen or positive HCV RNA (if necessary)
  4. History or evidence of well documented autoimmune hepatitis (i.e. specific autoantibodies, hypergammaglobulinemia, consistent histologic changes)
  5. History or evidence of primary biliary cholangitis (PBC)
  6. History or evidence of primary sclerosing cholangitis (PSC)
  7. History or evidence of Wilson's disease
  8. History or evidence of alpha-1-antitrypsin deficiency
  9. History or evidence of hemochromatosis
  10. History or evidence of drug-induced liver disease, as defined on the basis of typical exposure and history
  11. Known bile duct obstruction or a history of prior biliary tract diversion
  12. Suspected or proven liver cancer;
* History of human immunodeficiency virus (HIV) infection (positive HIV Ab);
* Patients with diabetes mellitus type 1;
* Patients with decompensated diabetes mellitus type 2 defined as either a HbA1c ≥ 9.5% at the time of screening or patients who are insulin dependent;
* Patients under evaluation for a suspected malignancy, with any history of hepatocellular carcinoma (HCC), or a history of other malignancy diagnosed or treated within 2 years prior to Randomization (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to Screening);
* Patients showing deleterious effects of alcohol abuse (as assessed by the investigator) or that consume excessive amounts of alcohol (>14 units/week for both females and males; for the purposes of this study one unit of alcohol is considered to be equal to 8 gr);
* Patients treated with chronic medication including but not limited to anti-retrovirals, tamoxifen, methotrexate, cyclophosphamide, isotretinoin, bile acid binding resins, obeticholic acid, ursodeoxycholic acid or pharmacologic doses of oral glucocorticoids (≥ 10 mg of prednisone per day or equivalent) within 12 weeks of Randomization
* Significant systemic or major illness other than liver disease including:

  1. Acute coronary syndrome, unstable angina, congestive heart failure, or cerebrovascular event within 24 weeks prior to Randomization
  2. Major surgery within 12 weeks prior to Randomization
  3. CNS disorders including Alzheimer's disease or other forms of dementia, seizure disorders and Parkinson's disease
  4. Autoimmune disease that has required systemic treatment in the 2 years preceding the study screening (i.e., with the use of disease-modifying agents, corticosteroids or immunosuppressive drugs)
  5. Uncontrolled thyroid disease
  6. Clinically significant renal dysfunction (estimated GFR < 60 ml/min (CKD equation))
  7. A history of any clinically significant medical disorder that, in the judgement of the investigator, would interfere with patient treatment, assessment, or compliance with the protocol;
* Known severe allergic or anaphylactic reactions to recombinant therapeutic proteins, fusion proteins, or chimeric, human, or humanized antibodies;
* Patients with any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing and protocol requirements.
* Participation in a study of another investigational agent within 28 days or five half-lives of the drug (whichever is longer) prior to screening;
* Prior treatment with CM-101 antibody

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Safety-related endpoints - Treatment emergent adverse events (TEAEs) | 14-week treatment period
  The safety and tolerability will be assessed by monitoring treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Serum biomarkers for pharmacodynamic parameters - Enhanced liver function (ELF™) Blood Test | Change from baseline to week 16
  Change in serum biomarkers for Enhanced liver function (ELF™) Blood Test
Serum biomarkers for pharmacodynamic parameters - Pro-C3 | Change from baseline to week 16
  Change in serum biomarkers for Pro-C3
Serum biomarkers for pharmacodynamic parameters - PRO-C4 | Change from baseline to week 16
  Change in serum biomarkers for PRO-C4
Serum biomarkers for pharmacodynamic parameters - C3M | Change from baseline to week 16
  Change in serum biomarkers for C3M
Serum biomarkers for pharmacodynamic parameters - Cytokeratin-18 (cCK-18) (full length and fragments; M65, M30) | Change from baseline to week 16
  Change in serum biomarkers for Cytokeratin-18 (cCK-18) (full length and fragments; M65, M30)
Serum inflammatory markers - Fibrinogen | From baseline over time
  Change over time in serum inflammatory markers - Fibrinogen
Serum inflammatory markers - C-reactive protein (CRP) | From baseline over time
  Change over time in serum inflammatory markers - C-reactive protein (CRP)
Change in liver enzymes | From baseline over time
  Absolute and percentage changes from Baseline over time through to week 16 as well as the percentage of normalization of ALT, AST, ALP, GGT, total bilirubin (TB) triglycerides and lipid profile (total cholesterol, HDL C, LDL C)
Immune cell sub populations evaluation | 16 weeks
  Whole Blood sampling for immune cell sub populations evaluation
Change in Liver Stiffness | Change from Baseline to week 16
  Change from Baseline to week 8 and 16 in liver stiffness using Transient Elastography
Change in Liver Fat Content | Change from Baseline to week 16
  Change from Baseline to week 8 and 16 in LFC (Liver fat content) assessed by MRI-PDFF
Change in liver fibrosis - Fibrosis-4 (FIB-4) score | 16 weeks
  Change from baseline to week 16 in: fibrosis-4 (FIB-4) score
Change in liver fibrosis - AST/ALT ratio | 16 weeks
  Change from baseline to week 16 in: AST/ALT ratio
Change in liver fibrosis -APRI (AST to platelet ratio index) | 16 weeks
  Change from baseline to week 16 in: APRI (AST to platelet ratio index)
Change in liver fibrosis -the Nonalcoholic fatty liver disease (NAFLD) Fibrosis Score | 16 weeks
  Change from baseline to week 16 in: the Nonalcoholic fatty liver disease (NAFLD) Fibrosis Score
Pharmacokinetics (PK) profile - Cmax | 14 weeks
  Elucidate CM-101 Serum PK profile - Observed maximum plasma concentration
Pharmacokinetics (PK) profile - Tmax | 14 weeks
  Elucidate CM-101 Serum PK profile - Time to reach the observed maximum plasma concentration (Cmax)
Pharmacokinetics (PK) profile - AUC∞ | 14 weeks
  Elucidate CM-101 Serum PK profile - Area under the plasma concentration-time curve extrapolated to infinity, calculated as: AUC∞ = AUClast + Clast/λz, where AUClast is the last measurable concentration.
Pharmacokinetics (PK) profile - t½ | 14 weeks
  Elucidate CM-101 Serum PK profile - Terminal elimination half-life, defined as 0.693/λz
Anti-Drug Antibodies | 14 weeks
  Evaluation of the development of anti-drug antibodies (ADA) following 14 weeks repeated administration

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frankel, MD, Study Director — ChemomAb Ltd.
Locations (9):
- Israel (9):
  - Soroka Medical Center - site 203, Beersheba
  - Carmel Medical Center - site 207, Haifa
  - Rambam Medical Center - site 202, Haifa
  - Hadassah Ein Kereme - site 201, Jerusalem
  - Shaare Zedek Medical Center - site 208, Jerusalem
  - Galilee Medical Center - site 204, Nahariya
  - Holy Family Nazareth Hospital - site 206, Nazareth
  - Rabin Medical Center - site 205, Petah Tikva
  - The Haim Sheba Medical Center - site 209, Ramat Gan

IPD SHARING:
Plan to Share IPD: No